CLINICAL TRIAL: NCT06031766
Title: Comparison of CIPA With the GLIM Criteria of Malnutrition and Prevalence of Sarcopenia in Inpatients
Brief Title: Comparison of CIPA With the GLIM Criteria and Prevalence of Sarcopenia in Inpatients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital of the Nuestra Señora de Candelaria (Other)
Responsible Party: Principal Investigator, Elena Marquez Mesa, Assistant doctor in Endocrinology and Nutrition, University Hospital of the Nuestra Señora de Candelaria
Other Study IDs: UniversityHNSC
Record Dates: First submitted 2023-08-20; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Malnutrition
Keywords: GLIM criteria; CIPA; phase angle; hospital stay; mortality; body composition; screening; Sarcopenia; inpatient; nutrition assessment
MeSH Terms: conditions — Malnutrition; Sarcopenia | interventions — Dietary Supplements

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Dietary supplement — The participation of the patients in the study will consist of performing the screening for malnutrition that is usually used in the hospital (CIPA) to which the GLIM test will be added, considered as the gold standard for this work. Subsequently, the sample of patients with a positive CIPA (as it is currently considered the screening test used in the hospital) will be implemented the therapeutic measures according to the usual protocol, while the subjects with a negative CIPA test but a positive GLIM will be studied. and constant monitoring taking the appropriate measures according to optional criteria. The patients will be followed up for the study of prognostic factors based on the variables obtained.

SUMMARY:
Determine the diagnostic quality of the CIPA tool, in inpatients with stays longer than three days, in the observation of risk of malnutrition compared to the gold standard GLIM as a diagnosis of malnutrition.

DETAILED DESCRIPTION:
Background: malnutrition is a poor prognostic factor in inpatients. Its early detection, together to nutritional intervention, can improve clinical evolution. It is important to carry out nutritional screening, however, there is no gold standard, and CIPA (Control of Intakes, Proteins and Anthropometry) has been implemented in our setting. The GLIM criteria (Global Leadership Initiative on Malnutrition) aim to provide a global consensus that allows common criteria for malnutrition diagnosis. The objective of this study is to evaluate the diagnostic quality of the CIPA screening vs the GLIM criteria for malnutrition as well as to establish the prevalence of sarcopenia.

Methods: cross-sectional single-center study comparing the diagnostic quality of CIPA in the diagnosis of malnutrition or risk of presenting it in inpatients vs GLIM. Adults of both sexes with a hospital stay of more than three days and attached to one of the following departments will be included: general surgery, internal medicine, vascular surgery, digestive system, hematology, nephrology, pulmonology, oncology, neurology, traumatology. The diagnostic evaluation of malnutrition and functionality will be carried out after three days of hospital stay, once the CIPA screening has been carried out. The participation of the patients in the study will consist of performing the CIPA malnutrition screening to which the GLIM test will be added. For the CIPA test, the BMI (body mass index), albumin levels and percentage of decreased intake will be taken. For the GLIM test, phenotypic criteria such as non-voluntary weight loss and reduction in muscle mass will also be studied together with etiological criteria to which, in addition to those referred to for the CIPA test, the presence of inflammation will be added. The study consists of a first cross-sectional part that will be completed once the data of the 490 subjects selected through probabilistic sampling has been collected. The second part of the study will consist of the prospective follow-up of the patients and the variables will be analyzed with prognostic criteria.

Discussion: this study will evaluate the diagnostic quality of CIPA vs the GLIM criteria for malnutrition and will establish the prevalence of sarcopenia in inpatients.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (> 18 years old).
* Hospital stay more than 3 days.
* Admitted to one of the following departments: general surgery, internal medicine, vascular surgery, digestive system, hematology, nephrology, pulmonology, oncology, neurology, traumatology.

Exclusion Criteria:

* Subjects with a prognosis of hospital stay less or equal than 3 days.
* Admitted to services with a low incidence of malnutrition: ophthalmology, dermatology or obstetrics.
* Admitted or critical care unit and palliative care.
* Pediatric patient.
* Patients treated with nutritional support before CIPA screening is performed.
* Patients with edema-ascitic overload.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects of both sexes with a hospital stay of more than three days.
Sampling Method: Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The concordance between CIPA test and the GLIM criteria determined by the Kappa coefficient. | 6 months

SECONDARY OUTCOMES:
Incidence of mortality | 6 months
Mean length of stay (days) | 6 months
Incidence of readmissions | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Elena Márquez Mesa, Physician, Principal Investigator — University HNSC
Locations (1):
- UniversityHNSC, Santa Cruz de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gomes F, Baumgartner A, Bounoure L, Bally M, Deutz NE, Greenwald JL, Stanga Z, Mueller B, Schuetz P. Association of Nutritional Support With Clinical Outcomes Among Medical Inpatients Who Are Malnourished or at Nutritional Risk: An Updated Systematic Review and Meta-analysis. JAMA Netw Open. 2019 Nov 1;2(11):e1915138. doi: 10.1001/jamanetworkopen.2019.15138. PMID 31747030
- [Result] Alvarez-Hernandez J, Planas Vila M, Leon-Sanz M, Garcia de Lorenzo A, Celaya-Perez S, Garcia-Lorda P, Araujo K, Sarto Guerri B; PREDyCES researchers. Prevalence and costs of malnutrition in hospitalized patients; the PREDyCES Study. Nutr Hosp. 2012 Jul-Aug;27(4):1049-59. doi: 10.3305/nh.2012.27.4.5986. PMID 23165541
- [Result] Zugasti Murillo A, Petrina-Jauregui ME, Ripa-Ciaurriz C, Sanchez Sanchez R, Villazon-Gonzalez F, Gonzalez-Diaz Faes A, Fernandez-Lopez C, Calles-Romero L, Martin Palmero MA, Riestra-Fernandez M, Dublang-Irazabal M, Rengel-Jimenez J, Diez-Muniz-Alique M, Agorreta-Ruiz JJ, Salsamendi-Perez JL, Larranaga-Unanue I, Abinzano-Guillen ML, Olariaga O, De la Cruz JJ. SeDREno study - prevalence of hospital malnutrition according to GLIM criteria, ten years after the PREDyCES study. Nutr Hosp. 2021 Oct 13;38(5):1016-1025. doi: 10.20960/nh.03638. PMID 34157845
- [Result] Mora Mendoza A, Suarez Llanos JP, Sanchez Morales A, Lorenzo Gonzalez C, Zambrano Huerta Y, Llorente Gomez de Segura I. Validation of CIPA nutritional screening through prognostic clinical variables in hospitalized surgical patients. Endocrinol Diabetes Nutr (Engl Ed). 2020 May;67(5):304-309. doi: 10.1016/j.endinu.2019.07.008. Epub 2019 Oct 24. English, Spanish. PMID 31668927
- [Result] Suarez Llanos JP, Benitez Brito N, Oliva Garcia JG, Pereyra-Garcia Castro F, Lopez Frias MA, Garcia Hernandez A, Diaz Sirgo B, Llorente Gomez de Segura I. [Introducing a mixed nutritional screening tool (CIPA) in a tertiary hospital]. Nutr Hosp. 2014 May 1;29(5):1149-53. doi: 10.3305/nh.2014.29.5.7299. Spanish. PMID 24951997
- [Result] Mendoza AM, Suarez Llanos JP, Delgado Brito I, Pereyra-Garcia Castro F, Lopez Travieso R, Perez Delgado N, Garcia Nunez MA, Benitez Brito N, Palacio Abizanda E. [Optimisation of nutritional screening tool CIPA: are two parameters of protein really necessary?]. Nutr Hosp. 2018 Aug 2;35(4):914-919. doi: 10.20960/nh.1701. Spanish. PMID 30070882
- [Result] Suarez-Llanos JP, Mora-Mendoza A, Benitez-Brito N, Perez-Mendez L, Pereyra-Garcia-Castro F, Oliva-Garcia JG, Palacio-Abizanda JE. Validity of the new nutrition screening tool Control of Food Intake, Protein, and Anthropometry (CIPA) in non-surgical inpatients. Arch Med Sci. 2018 Aug;14(5):1020-1024. doi: 10.5114/aoms.2017.66084. Epub 2017 Feb 20. PMID 30154883
- [Result] Suarez-Llanos JP, Vallejo-Torres L, Garcia-Bello MA, Hernandez-Carballo C, Calderon-Ledezma EM, Rosat-Rodrigo A, Delgado-Brito I, Pereyra-Garcia-Castro F, Benitez-Brito N, Felipe-Perez N, Ramallo-Farina Y, Romero-Perez JC. Cost-effectiveness of the hospital nutrition screening tool CIPA. Arch Med Sci. 2019 Jan 11;16(2):273-281. doi: 10.5114/aoms.2018.81128. eCollection 2020. PMID 32190136
- [Result] Suarez-Llanos JP, Benitez-Brito N, Vallejo-Torres L, Delgado-Brito I, Rosat-Rodrigo A, Hernandez-Carballo C, Ramallo-Farina Y, Pereyra-Garcia-Castro F, Carlos-Romero J, Felipe-Perez N, Garcia-Niebla J, Calderon-Ledezma EM, Gonzalez-Melian TJ, Llorente-Gomez de Segura I, Barrera-Gomez MA. Clinical and cost-effectiveness analysis of early detection of patients at nutrition risk during their hospital stay through the new screening method CIPA: a study protocol. BMC Health Serv Res. 2017 Apr 20;17(1):292. doi: 10.1186/s12913-017-2218-z. PMID 28424063
- [Result] Cederholm T, Jensen GL, Correia MITD, Gonzalez MC, Fukushima R, Higashiguchi T, Baptista G, Barazzoni R, Blaauw R, Coats A, Crivelli A, Evans DC, Gramlich L, Fuchs-Tarlovsky V, Keller H, Llido L, Malone A, Mogensen KM, Morley JE, Muscaritoli M, Nyulasi I, Pirlich M, Pisprasert V, de van der Schueren MAE, Siltharm S, Singer P, Tappenden K, Velasco N, Waitzberg D, Yamwong P, Yu J, Van Gossum A, Compher C; GLIM Core Leadership Committee; GLIM Working Group. GLIM criteria for the diagnosis of malnutrition - A consensus report from the global clinical nutrition community. Clin Nutr. 2019 Feb;38(1):1-9. doi: 10.1016/j.clnu.2018.08.002. Epub 2018 Sep 3. PMID 30181091
- [Result] Correia MITD, Tappenden KA, Malone A, Prado CM, Evans DC, Sauer AC, Hegazi R, Gramlich L. Utilization and validation of the Global Leadership Initiative on Malnutrition (GLIM): A scoping review. Clin Nutr. 2022 Mar;41(3):687-697. doi: 10.1016/j.clnu.2022.01.018. Epub 2022 Feb 1. PMID 35151125
- [Result] Garlini LM, Alves FD, Ceretta LB, Perry IS, Souza GC, Clausell NO. Phase angle and mortality: a systematic review. Eur J Clin Nutr. 2019 Apr;73(4):495-508. doi: 10.1038/s41430-018-0159-1. Epub 2018 Apr 26. PMID 29695763
- [Result] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jul 1;48(4):601. doi: 10.1093/ageing/afz046. No abstract available. PMID 31081853
- [Result] Boulhosa RSSB, Lourenco RP, Cortes DM, Oliveira LPM, Lyra AC, de Jesus RP. Comparison between criteria for diagnosing malnutrition in patients with advanced chronic liver disease: GLIM group proposal versus different nutritional screening tools. J Hum Nutr Diet. 2020 Dec;33(6):862-868. doi: 10.1111/jhn.12759. Epub 2020 May 7. PMID 32378264
- [Result] Clark AB, Reijnierse EM, Lim WK, Maier AB. Prevalence of malnutrition comparing the GLIM criteria, ESPEN definition and MST malnutrition risk in geriatric rehabilitation patients: RESORT. Clin Nutr. 2020 Nov;39(11):3504-3511. doi: 10.1016/j.clnu.2020.03.015. Epub 2020 Mar 23. PMID 32273200
- [Result] Bellanti F, Lo Buglio A, Quiete S, Pellegrino G, Dobrakowski M, Kasperczyk A, Kasperczyk S, Vendemiale G. Comparison of Three Nutritional Screening Tools with the New Glim Criteria for Malnutrition and Association with Sarcopenia in Hospitalized Older Patients. J Clin Med. 2020 Jun 17;9(6):1898. doi: 10.3390/jcm9061898. PMID 32560480
- [Result] Ballesteros-Pomar MD, Gajete-Martin LM, Pintor-de-la-Maza B, Gonzalez-Arnaiz E, Gonzalez-Roza L, Garcia-Perez MP, Gonzalez-Alonso V, Garcia-Gonzalez MA, de Prado-Espinosa R, Cuevas MJ, Fernandez-Perez E, Mostaza-Fernandez JL, Cano-Rodriguez I. Disease-Related Malnutrition and Sarcopenia Predict Worse Outcome in Medical Inpatients: A Cohort Study. Nutrients. 2021 Aug 25;13(9):2937. doi: 10.3390/nu13092937. PMID 34578815
- [Result] Lengele L, Bruyere O, Beaudart C, Reginster JY, Locquet M. Malnutrition, assessed by the Global Leadership Initiative on Malnutrition (GLIM) criteria but not by the mini nutritional assessment (MNA), predicts the incidence of sarcopenia over a 5-year in the SarcoPhAge cohort. Aging Clin Exp Res. 2021 Jun;33(6):1507-1517. doi: 10.1007/s40520-021-01880-5. Epub 2021 May 15. PMID 33991331

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT06031766/Prot_SAP_000.pdf